CLINICAL TRIAL: NCT06369623
Title: Neuromelanin MRI: A Tool for Non-invasive Investigation of Dopaminergic Abnormalities in Adolescent Substance Use
Brief Title: Monetary Incentive Delay Task for Probing Reward-related Neural Processes
Acronym: MID
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Greg Perlman, Principal Investigator, Stony Brook University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB2023-00466
Record Dates: First submitted 2024-04-13; First posted 2024-04-17 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Adolescent Development

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Whole sample (Experimental): All enrolled subjects will complete a standard Monetary Incentive Delay Task if able. Inclusion of this task meets criteria for Basic Experimental Studies Involving Humans (BESH)
  Interventions: Other: Monetary Incentive Delay Task

INTERVENTIONS:
Other: Monetary Incentive Delay Task — The Monetary Incentive Delay functional Magnetic Resonance Imaging task is well-characterized and commonly utilized in research settings to measure neural activation between win and loss conditions, as well as between phases of anticipation and consummation/outcome. A recent meta-analysis indicates that the task has been used in over 80 studies and 5,000 subjects as of Year 2022. The task is also valid and appropriate for use in children and adolescents, as demonstrated by its inclusion in National Institute on Drug Abuse ABCD study. The task is utilized for its short-lived, reversible, and/or benign effects on brain activation (e.g., brief processing of a reward cue).

SUMMARY:
150 males and 150 females ages 14-17 years-old will be enrolled in an observational, longitudinal study. There are three planned in-person visits: a baseline assessment, an 18-month follow-up, and a 36-month follow-up. The in-person visits will include assessment of substance use and other individual differences (e.g., reward function, psychiatric history), neuromelanin-sensitive MRI, as well as functional brain activation collected while the participant is at rest (resting-state fMRI) and while the participant completes a Monetary Incentive Delay task. Subjects will also be asked to complete past 90-day substance use assessments remotely every 90 days for 36 months.

DETAILED DESCRIPTION:
Substance use disorders affect several million people in the United States every year, create significant economic burden, and cause tremendous suffering at the person, family, and societal levels. This proposal aims to investigate the dynamic interplay between pediatric substance use (a risk factor for substance use disorders) and rate of neuromelanin accumulation (a proxy for dopamine function) for the first time. Thus, this research seeks to identify a brain mechanism (dopamine function) that could be targeted in youth by future treatments in order to prevent onset of substance use disorders.

The goals of this study require a prospective imaging design that relies on the naturally-occurring adolescent substance use (e.g., differences in timing and amount of substance use is treated as quasi-experimental). Importantly, the investigators will begin data collection in a cohort on the cusp of entering a high-risk period of substance use initiation and conclude data collection after 36-months to capture substance use escalation. An intermediate 18-month follow-up NM-MRI scan is needed to help clarify the magnitude of early changes in NM accumulation. Thus, this is a longitudinal, observational study.

Of note, the use of the Monetary Incentive Delay fMRI task at baseline, 18-month, and 36-month follow-ups fulfills the NIH criteria of a basic experimental studies involving humans (BESH). Thus, this study as a whole qualifies as a clinical trial based on the determination:

1. The study involves humans
2. The participants are prospectively assigned to an intervention, which in this case means that the subject will be assigned to complete the Monetary Incentive Delay fMRI task while lying in the MRI scanner.
3. The study is designed to evaluate the effect of the intervention on participants, which in this case means that the investigators will evaluate the effect of the Monetary Incentive Delay task on brain activation in participants.
4. The effect being evaluated is a health-related biomedical or behavioral outcome, which in this case means fMRI brain activation between win and loss conditions, as well as between phases of anticipation and consummation/outcome.

In brief, use of this fMRI task is a single arm, non-masked, non-randomized, basic science intervention. This does not match any of the NIH-defined clinical trials phases (n/a). The fMRI data (brain activation) is the primary outcome measure of the BESH intervention, but is a tertiary outcome in the context of this longitudinal study. The task is utilized for its short-lived, reversible, and benign effects (e.g., brief changes in brain activation).

ELIGIBILITY:
Inclusion Criteria:

* Males and females ages 14-17 years-old;
* English-speaking for assent and interview completion;
* Capacity to provide assent.
* For parents, the inclusion criteria will be willing and capacity to provide parental permission/consent.

Exclusion Criteria:

* current (within 6 months) use of medication that may affect cerebral function
* history of severe medical or neurological illness, including stroke or seizure;
* history of head trauma with loss of consciousness;
* presence of metal in the body;
* pregnancy or breastfeeding;
* recent drug or alcohol use determined by positive urine toxicology or breathalyzer (to validate self-report assessment of substance use history);
* lifetime use of psychotropic or other medication that could likely influence dopamine function, namely stimulant medication or antipsychotic medication, except a subgroup of 25 youth with history of prescribed stimulant medication and a subgroup of 15 youth with history antipsychotic medication will be enrolled for comparison purposes.

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2024-04-06 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Amount of Brain Activation (BOLD Signal) during Monetary Incentive Delay Task by Condition | Baseline, 18-month, 36-month.
  fMRI activation during task during win, loss, and no change conditions, as well as anticipation and consummation phases.

CONTACTS AND LOCATIONS:
Locations (1):
- Stony Brook Medicine, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No